CLINICAL TRIAL: NCT00541593
Title: Natural Orifice Translumenal Endoscopic Surgery (NOTES) Cystgastrostomy for the Treatment of Pancreatic Pseudocysts
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: SurgAssist device is no longer clinically available.
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, John Romanelli, Medical Director, Weight Loss Surgery Program, Baystate Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-164
Record Dates: First submitted 2007-10-07; First posted 2007-10-10 (Estimated); Results first posted 2013-11-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-09

CONDITIONS: Pancreatic Pseudocyst
Keywords: Pancreatic pseudocyst; NOTES
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NOTES pancreatic pseudocystgastrostomy (Experimental): Patients who undergo pancreatic pseudocystgastrostomy via a NOTES technique.
  Interventions: Procedure: Pancreatic Pseudocystgastrostomy

INTERVENTIONS:
Procedure: Pancreatic Pseudocystgastrostomy — An operation to connect the pancreatic pseudocyst to the stomach so it can drain into the stomach and intestines

SUMMARY:
Natural Orifice Translumenal Endoscopic Surgery (NOTES) describes a new field of investigational surgery which uses the endoscope as the primary operative tool. The insertion sites for the endoscope include natural orifices such as the mouth, anus, vagina, or urethra. Multidisciplinary teams consist of surgeons and gastroenterologists who are collaborating to develop safe and effective surgical techniques via the natural orifice route in order to avoid surgical incisions. Pancreatic pseudocysts are cavities that form typically in the lesser sac following an episode of acute pancreatitis, that may be able to be drained by a variety of techniques, including endoscopically. Chronic pseudocysts often require surgical drainage into the stomach. The medical device company known as "Power Medical Interventions" has a computer-powered surgical stapler which rests on a flexible shaft. Following the insertion of the endoscope, the powered stapler will be passed alongside the endoscope to help the surgeon and gastroenterologist (working as a team) to see where to properly place the stapler. Once the stapler is in position, one jaw of the stapler will be placed into the pseudocyst, and the other jaw will be left in the stomach. The stapler will then be closed and fired, creating a permanent connection between the two hollow spaces and allow the contents of the pseudocyst to drain naturally out into the stomach and intestines. Utilizing this technique, a surgical incision is avoided.

Hypothesis: Patients who undergo the Natural Orifice Translumenal Endoscopic Surgery for treatment of their pancreatic pseudocyst will experience effective treatment with less discomfort and with quicker recovery than standard surgical techniques.

DETAILED DESCRIPTION:
Introduction: Natural Orifice Translumenal Endoscopic Surgery (NOTES) describes a new field of investigational surgery which uses the endoscope as the primary operative tool. Multiple animal studies utilizing similar techniques are ongoing at several institutions, including Baystate Medical Center. These multidisciplinary teams consist of surgeons and gastroenterologists who are collaborating to develop safe and effective surgical techniques via the natural orifice route in order to avoid surgical incisions.

Pancreatic pseudocysts are cavities that form typically in the lesser sac following an episode of acute pancreatitis. These pseudocysts may become infected, and may have detrimental outcomes caused by their mass effect on the stomach and/or small intestine. Pseudocysts are able to be drained by a variety of techniques, including endoscopically. Chronic pseudocysts often require surgical drainage into the stomach or jejunum as they may contain solid material that does not drain. Typically, cystgastrostomies or cystenterotomies are performed utilizing an abdominal incision with subsequent suturing or stapling.

The medical device company known as "Power Medical Interventions" has a computer-powered surgical stapler which rests on a flexible shaft. There has been subsequent development of a linear version of this stapler which was designed for gastrointestinal anastomosis which will be utilized in this research project known as a "powered stapler".

An endoscope would be inserted in the mouth, and down into the stomach after the induction of general anesthesia. Following the insertion of the endoscope, the powered stapler will be passed alongside the endoscope to help the surgeon and gastroenterologist (working as a team) to see where to properly place the stapler. If a connection has been previously made between the stomach and pseudocyst, the stapler will be maneuvered into the proper position. If a connection has not yet been made, this will be done during the procedure with the aid of an endoscopic ultrasound probe passed through the mouth. Once the stapler is in position, one jaw of the stapler will be placed into the pseudocyst, and the other jaw will be left in the stomach. The stapler will then be closed and fired, creating a permanent connection between the two hollow spaces and allow the contents of the pseudocyst to drain naturally out into the stomach and intestines. The stapler and the endoscope are then removed and the anesthesia is allowed to wear off. Utilizing this technique, a surgical incision is avoided.

Primary Objective: The primary objective of this study is to demonstrate that the Natural Orifice Translumenal Endoscopic Surgery (NOTES) technique is as effective as standard surgical technique for the permanent drainage of pancreatic pseudocysts.

Secondary Objective: The secondary objective of this research project is to demonstrate a decreased degree of pain experienced by patients undergoing the Natural Orifice Translumenal Endoscopic Surgery versus traditional methods.

Hypothesis: Patients who undergo the Natural Orifice Translumenal Endoscopic Surgery for treatment of their pancreatic pseudocyst will experience effective treatment with less discomfort and with quicker recovery than standard surgical techniques.

Background: The NOTES team (surgeon and gastroenterologist) at Baystate has extensive experience with animal work in developing novel techniques with commercially available products. While we have not ever performed a cystgastrostomy on an animal, there is no known animal model to simulate this pathologic condition. We have, however, operated the flexible gastrointestinal anastomotic stapler translumenally in an animal model in order to prepare for this procedure. The surgeon on the team has performed human stapled cystgastrostomies before, via both open and laparoscopic approaches. A pilot case has recently been done performed and the patient continues to do well.

Study Design: There will be a total of 10 patients undergoing this experimental surgical procedure once meeting all entry criteria and subsequent to obtaining informed consent. Follow-up endoscopic examination will be conducted approximately 6 weeks following the procedure to determine the success of the drainage of the pseudocyst. Longer term follow-up will be determined by the patient's overall condition. These 10 patients will be compared to a retrospective review of 10 patients to compare pseudocyst size, degree of pain and hospital length of stay. The degree of pain will be assessed using the Wong-Baker Pain Scale. The retrospective series will be a matched cohort based on size of the pseudocyst and age and comorbidities of the patient.

Safety Monitoring: Due to the novelty of the procedure, safety information will be monitored on a continuous basis. Should there be any untoward results, the study may be terminated prematurely, or temporarily suspended while we assess the events. In the event of any serious adverse event or outcome, the IRB will be notified immediately.

Risks and Benefits: The anticipated risks associated with this type of surgery include:

Bleeding, infection, need for open surgery, pancreatic leak, gastric leak, inadequate drainage of the pseudocyst. A risk specific to the NOTES approach includes trauma to oropharynx resulting in bleeding or infection.

The anticipated benefits include a decrease in the amount of pain experienced with the drainage of the pancreatic pseudocyst, as well as an anticipated decreased length of hospital stay.

Statistics: A comparison of the means will be performed using both the numerical values from the Pain Scale, the largest diameter of the pseudocyst, and the hospital length of stay.

Data Storage: The data collected will be kept in a locked filing cabinet in the primary investigator's office. Only the PI will have access to this file.

Enrollment Inclusion Criteria:

1. Adult (over 18 years old) patients who are able to provide informed consent for this surgical procedure
2. Patients scheduled to undergo non-emergent surgical treatment removal of pancreatic pseudocyst

Enrollment Exclusion Criteria:

1. Inability to provide informed consent
2. Patients who, in the opinion of the investigator, would not be appropriate for enrollment into this experimental research project
3. Patients who are deemed to be unstable from a medical standpoint to undergo pancreatic surgery
4. Pregnancy

It is anticipated that there will be more similar type of "natural orifice" type surgeries in the future for a variety of procedures and a multitude of reasons (no incision, less pain, and less time in the hospital). This surgery is the first of its kind for the drainage of pancreatic pseudocysts.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (over 18 years old) patients who are able to provide informed consent for this surgical procedure
2. Patients scheduled to undergo non-emergent surgical treatment removal of pancreatic pseudocyst

Exclusion Criteria:

1. Inability to provide informed consent
2. Patients who, in the opinion of the investigator, would not be appropriate for enrollment into this experimental research project
3. Patients who are deemed to be unstable from a medical standpoint to undergo pancreatic surgery
4. Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-09; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Romanelli, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NOTES Pancreatic Pseudocystgastrostomy Patients: Patients who undergo pancreatic pseudocystgastrostomy via a NOTES technique. All of them are candidates for open or laparoscopic pancreatic pseudocystgastrostomy, but have chosen a less invasive result. Also, all of them have to have imaging criteria which suggest that the stomach and pseudocyst are in close contact, and that the cyst is proximal enough in the stomach to be reachable with an endoscope and/or endoscopic stapler.
Period: Overall Study
Arm/Group | NOTES Pancreatic Pseudocystgastrostomy Patients
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NOTES Pancreatic Pseudocystgastrostomy Patients
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 55.8 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Number of patients who died as a result of the surgery: Death (mortality).
  Please note that pain was previously listed as an outcome measure, but this was edited out of this submission and was not tracked as an outcome measure.
Time Frame: One year
Population: Patients who had the diagnosis, qualified anatomically, and were interested in the research study (and who met inclusion criteria but not exclusion criteria) were enrolled.
Measure: Number; unit: participants
Groups:
- NOTES Pancreatic Pseudocystgastrostomy Patients: Pancreatic Pseudocystgastrostomy Patients having NOTES procedure
Arm/Group | NOTES Pancreatic Pseudocystgastrostomy Patients
Number analyzed (Participants) | 5
participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | NOTES Pancreatic Pseudocystgastrostomy Patients
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Early termination due to the company that made the device going out of business; the company that acquired it chose not to market the device. Given the lack of clinical support, we chose to terminate the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes